CLINICAL TRIAL: NCT04102319
Title: Association Between Hepcidin, Haemoglobin Level and Iron Status in Stage 4 Chronic Kidney Disease Patients With Anaemia
Brief Title: Serum Hepcidin, Haemoglobin Level and Iron Status in Chronic Kidney Disease Patients (CKD) With Anaemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Deiaaeldeen Masaoud Sadeq Mohammed, Dr, Assiut University
Other Study IDs: hepcidin,Anemia
Record Dates: First submitted 2019-09-19; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: CKD Stage 4

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum hepcidin — it is a serum marker

SUMMARY:
The current study is planned to assess possible relationships of serum hepcidin levels with haemoglobin levels, inflammation and iron statuses in stage 4 CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years) with anaemia who had CKD stage 4 with glomerular filtration rate (GFR) 15-29 ml/min/1.73 m2

Exclusion Criteria:

* Subjects with blood transfusion within the preceding 3 months. myocardial infarction (MI) history within the preceding 3 months, surgical history within the preceding 3 months, malignancy. Advanced liver cirrhosis. uncontrolled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic kidney disease stage 4 who have anemia with hemoglobin level below 11 gm/dl
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
relation between serum hepcidin level and ESR ckd stage 4 | at study entry and then again after 3 months
  measure strength of relation, r, between levels of serum hepcidin and ESR, an inflammation marker
relation between serum hepcidin and serum ferritin levels | at study entry and then again after 3 months
  measure strength of relation, r, between levels of hecidin and ferritin

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hamed, MD, Principal Investigator — Assiut University